CLINICAL TRIAL: NCT00066456
Title: A Phase I Study Using Low Dose Abdominal Radiotherapy as A Docetaxel Chemosensitizer for Recurrent , Persistent Or Advanced Ovarian, Peritoneal Or Fallopian Tube Cancer
Brief Title: Radiation Therapy to the Abdomen Plus Docetaxel in Treating Patients With Recurrent or Persistent Advanced Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9915; NCI-2009-00618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000316238; GOG-9915; GOG-9915 (Other: Gynecologic Oncology Group); GOG-9915 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Recurrent Ovarian Carcinoma; Stage III Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Radiotherapy, Conformal; Docetaxel

ARMS (1):
- Treatment (chemosensitization, radiation, docetaxel) (Experimental): Patients receive docetaxel IV over 30 minutes once daily on days 1, 8, 15, 22, 29, and 35. Within 3 hours after beginning docetaxel, patients also receive low-dose abdominal radiotherapy twice daily (at least 4 hours apart) on days 1, 2, 8, 9, 15, 16, 22, 24, 29, 30, 35, and 36. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Chemosensitization/Potentiation Therapy; Drug: Docetaxel

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Chemosensitization/Potentiation Therapy
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate

SUMMARY:
Phase I trial to study the effectiveness of low-dose radiation therapy to the abdomen combined with docetaxel in treating patients who have recurrent or persistent advanced ovarian, peritoneal, or fallopian tube cancer. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of docetaxel in combination with low-dose abdominal radiotherapy in patients with recurrent or persistent advanced ovarian, peritoneal, or fallopian tube cancer.

II. Determine the safety and toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of docetaxel.

Patients receive docetaxel IV over 30 minutes once daily on days 1, 8, 15, 22, 29, and 35. Within 3 hours after beginning docetaxel, patients also receive low-dose abdominal radiotherapy twice daily (at least 4 hours apart) on days 1, 2, 8, 9, 15, 16, 22, 24, 29, 30, 35, and 36. Treatment continues in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian, peritoneal, or fallopian tube carcinoma
* Radiographic, clinical, or pathologic evidence of relapse
* Recurrent or persistent disease after chemotherapy (may be enrolled at first or subsequent relapse)

  * Received prior taxane OR platinum agent
* Performance status - GOG 0-1
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No grade 2 or greater neuropathy (sensory or motor)
* No septicemia
* No severe infection
* No circumstance that would preclude study completion
* No prior radiotherapy to the abdomen or pelvis
* Patients with ureteral obstruction must undergo stent or nephrostomy tube replacement prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-09; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Incidence of acute toxicity, graded using Common Toxicity Criteria version 2.0 | Up to 30 days after completion of radiation therapy

SECONDARY OUTCOMES:
Incidence of patients with chronic toxicity assessed by Common Toxicity Criteria version 2.0 Radiation Therapy Oncology Group/European Organization for Research and Treatment of Cancer (CTC v2.0 RTOG/EORTC) late radiation morbidity scoring | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fracasso, Principal Investigator — Gynecologic Oncology Group
Locations (7):
- United States (7):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Case Western Reserve University, Cleveland, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma